CLINICAL TRIAL: NCT02573142
Title: A Novel Healthcare-Community Partnership for Childhood Obesity Treatment: A Randomized Pilot Study
Brief Title: Integrated Child Obesity Treatment Study: Bull City Healthy and Fit
Acronym: BCHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066366
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Childhood Obesity
Keywords: obesity; treatment; community; integrated
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education-only (Active Comparator): Subjects in the education-only control will receive standard of care clinical treatment in the Duke Healthy Lifestyles clinic and educational materials describing community-based resources for physical activity and how to access them.
  Interventions: Behavioral: Healthy Lifestyles Clinic
- Bull City Fit Intervention (Experimental): Subjects in the Bull City Fit intervention will receive standard of care clinical treatment in the Duke Healthy Lifestyles clinic and unlimited access to a community-based wellness program that includes physical fitness activities and cooking classes.
  Interventions: Behavioral: Bull City Healthy and Fit

INTERVENTIONS:
Behavioral: Bull City Healthy and Fit — Integrated model of child obesity treatment including clinical care plus community-based program for family-based experiential learning of healthy habits.
  Arms: Bull City Fit Intervention
Behavioral: Healthy Lifestyles Clinic — Clinic-only model of care including clinical care and educational materials
  Arms: Education-only

SUMMARY:
The primary aim of this study is to reduce body mass index (BMI) among children ages 5-11 who are obese by integrating behavioral treatment strategies in both clinic (Healthy Lifestyles) and community (Bull City Fit) settings. A two-group randomized, controlled, non-blinded pilot design will be utilized. The intended target population is the adult caregiver and a child with obesity (BMI ≥ 95th percentile) aged 5-11. The intervention condition will be standard care with Healthy Lifestyles programming plus Bull City Fit; upcoming activities will be texted to the parents mobile device using GoogleVoice. The control condition will be standard clinical care with Healthy Lifestyles programming. Primary outcome is BMI at 6 months. Secondary outcomes include anthropometric, psychosocial, and reported health behaviors.

DETAILED DESCRIPTION:
Prevention strategies have made important strides to stabilize obesity prevalence, however US childhood obesity prevalence remains high (17%) and effective treatment has been elusive. Furthermore, children with severe obesity continues to increase, especially among Hispanics and African Americans. These children have increased cardio-metabolic risks and comorbidities, and healthcare costs are concentrated among them. It is critical to identify effective interventions that can be made widely available for low-income, diverse populations in order to mitigate economic and societal costs.

High-intensity behavioral treatment interventions in specialized clinical research settings have been shown to be modestly effective.Effects tend to be small, short-term, and difficult to replicate in "real-world" clinical settings. Community-based settings (e.g., recreation centers) offer an attractive setting to deliver treatment. Community centers are locally accessible, can offer activities during evenings and on weekends, and provide relaxed environments that support social interaction. However, community-based interventions cannot provide the patient-centered medical care and individual nutrition counseling currently recommended for obesity treatment. New recommendations encourage linking clinical treatment with community resources, yet evidence demonstrating the feasibility and efficacy of such interventions is limited.

Locally, the investigators have developed both a specialized clinical obesity treatment program as well as a community based treatment program, and have linked the two via a shared use agreement. The innovative model provides multidisciplinary, individualized behavioral modification counseling and support through the clinic-based Healthy Lifestyles program, and higher intensity social and environmental support to reinforce behavior change through Bull City Fit programming.

The clinical program, Duke Children's Healthy Lifestyles (HL), is a comprehensive (AAP Stage 2-4) childhood obesity treatment program that has served primarily low-income African American and Hispanic families since 2006. In short, children aged 22 years and under with BMI ≥ 95th percentile (i.e., obese) are referred by their primary physician to the multidisciplinary Healthy Lifestyles clinic for treatment of obesity and related co-morbidities. The intervention involves monthly visits for one year to meet with medical, dietary, exercise and behavior specialists all certified in Motivational Interviewing. Similar to other interventions delivered through primary care settings, the Healthy Lifestyles model alone leads to measurable but not clinically significant decreases in body mass index.

The community-based program, Bull City Fit (BCF), was developed in 2012 by HL staff to increase intensity of the clinical intervention. The community center is a Durham Parks and Recreation (PR) facility. The investigators chose this municipal partner due to potential scalability of the intervention; over 5,000 PR facilities exist nationwide and every American lives within a 20 mile radius of a PR facility (DPR.gov). Bull City Fit provides free access to Edison Johnson Community Center, including 2 hours of staffed programming six days a week designed specifically for Healthy Lifestyles patients aged 2-18 and their families. This includes sports, games, cooking classes, gardening, parent support groups, teen support groups, and developmentally appropriate activities for all ages. With guidance from Healthy Lifestyles clinic providers, Bull City Fit programming is run by trained volunteers who are primarily Duke University students, pediatric residents, and community members invested in the wellness of families in their city.

New treatment models with potential for both scalability and effect are critically needed to defray the estimated $14.1 billion annual direct costs of childhood obesity (e.g., prescription drugs, emergency and outpatient visits),5 which will only rise substantially as children with obesity become adults with obesity. The healthcare-community partnership model has been operational since 2012, primarily reaching a low-income and racially diverse population. The model has potential to scale via establishment of similar partnerships in other communities. The goal of the present study is to provide important new information about the effectiveness of the model, which can be used to refine and tailor the intervention for future expansion.

Study interventions

Trained clinical providers will collect and perform assessments that are in accordance with the current clinical protocol. A trained research assistant will collect all other measures either through chart review or direct questioning of the parent and/or child. Subjects will be randomized to the intervention or control group using a random number generator (Excel, 2010). A sample of 10 subjects will receive an accelerometer for 1 week as described above.

Subjects randomized to the standard care control group includes a lifestyle counseling visit, educational materials, goal-setting by a physician and dietician, and information about general community parks and recreation resources. After 6 months, control participants will receive invitation to participate in Bull City Fit. Subjects randomized to the intervention group will receive standard care as above plus invitation to participate in Bull City Fit. During the initial Healthy Lifestyle clinic appointment, the intervention participants will receive an introductory packet of information about Bull City Fit, and both the clinical providers and the research assistant will discuss the program verbally with the parent and child. The parent will be instructed to attend their first Bull City Fit session the Saturday subsequent to their clinical appointment, during which they will receive an orientation to the program and complete contracts that specify ground rules for the sessions (e.g., adult caregiver must accompany their child patient, cell phones are not allowed except for emergencies, etc.) and their commitment to actively participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 or older and is the child's primary caregiver ("parent")
* Child aged 5-11 years
* Child with age- and gender-specific BMI ≥ 95th percentile

Exclusion Criteria:

* Inability to read and write in English
* Family currently has paid membership to a gym or fitness center
* Parent with severe medical or mental health condition limiting ability to attend appointments
* Child with severe medical or mental health condition limiting ability to attend appointments or participate in behavioral therapies
* Parent and child live greater than 30 miles from the Duke Healthy Lifestyles clinic
* Plan to move out of state in next 6 months
* Child with medical condition as cause of obesity (e.g., hypothyroidism, Cushing's Syndrome, Prader-Willi syndrome (PWS), drug-induced obesity)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | 3 and 6 months
  Body mass index will be measured at 3- and 6-months post-enrollment.

SECONDARY OUTCOMES:
Change in Health habits | 3- and 6-month
  Self-reported fruit and vegetable consumption, and sugary drink consumption at 3 and 6 months post-intervention
Change in Cardiovascular fitness | 3- and 6-months
  Score on 3-minute step test at 3- and 6-months post-enrollment
Change in Adherence to clinic appointments | 3- and 6- months
  Number of clinic appointments patient attended at 3- and 6-months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke Children's Health Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hoffman J, Frerichs L, Story M, Jones J, Gaskin K, Apple A, Skinner A, Armstrong S. An Integrated Clinic-Community Partnership for Child Obesity Treatment: A Randomized Pilot Trial. Pediatrics. 2018 Jan;141(1):e20171444. doi: 10.1542/peds.2017-1444. Epub 2017 Dec 13. PMID 29237800